CLINICAL TRIAL: NCT01797627
Title: Ventricular Size Involvement in Neuropsychological Outcomes in Pediatric Hydrocephalus (VINOH)
Brief Title: Ventricular Size Involvement in Neuropsychological Outcomes in Pediatric Hydrocephalus
Acronym: VINOH
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Hydrocephalus Association (Other)
Responsible Party: Principal Investigator, richard holubkov, Ph.D., University of Utah
Other Study IDs: 49237; 1RC1NS068943-01 (NIH); HCRN 006 (Other: HCRN Protocol Number)
Record Dates: First submitted 2012-06-08; First posted 2013-02-22 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Hydrocephalus
Keywords: Pediatric Hydrocephalus; Ventricular Size; Neuropsychological Outcomes; Quality of Life
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This multicenter, prospective study of children with hydrocephalus will examine whether or not ventricle size is associated with poor cognitive outcomes. It is expected that results will indicate larger ventricular size at 6 months after surgery for the initial treatment of hydrocephalus will relate to poorer cognitive outcomes. This study is being conducted by the Hydrocephalus Clinical Research Network (HCRN), a network established to conduct multi-institutional clinical trials on pediatric hydrocephalus.

DETAILED DESCRIPTION:
The current literature is inconclusive regarding the direct association between large ventricle size and poorer cognitive outcomes. This uncertainty stems from relatively few studies, problems with study design (possible confounding factors), varying study populations of hydrocephalus, and conflicting evidence. If the association is proven then aggressive strategies must be developed to maximally decrease ventricular size in these children to preserve long-term cognitive functioning. However, if the association is disproven then previous reservations for procedures such as Endoscopic Third Ventriculostomy (ETV) or higher-resistance shunting to prevent overdrainage complications will be further minimized. Either finding has a major potential to further improve the quality of life in our pediatric hydrocephalus patients. This study is unique as it will include pediatric patients presenting with hydrocephalus from a wide range of etiologies. This study is also unique in that we propose to conduct a brief pre-operative neuropsychological examination to act as internal controls along with the outcomes obtained at a more extensive neuropsychological examination at six months after initial hydrocephalus treatment surgery.

ELIGIBILITY:
Inclusion Criteria: Patients will be eligible for enrollment if they:

* are 5 years of age or older; and
* have been newly diagnosed with hydrocephalus to be managed surgically with either a cerebrospinal fluid (CSF) shunt or an ETV; and
* have one of the following etiologies for hydrocephalus: aqueductal stenosis, supratentorial and posterior fossa tumors both benign and malignant, post-traumatic, myelomeningocele, tectal gliomas, post-infectious, and following spontaneous intraventricular hemorrhage (IVH). Malignant tumors have been included as the neuropsychological deficits secondary to adjuvant chemotherapy and radiation have not been demonstrated within the proposed study's 6 month window.

Exclusion Criteria: Patients will be ineligible for enrollment if ANY of the following is true or anticipated:

* present with a Glasgow Coma Scale (GCS) score of less than 14/15, cerebellar mutism, or cognitive deficits so severe as to make neuropsychological testing impossible; OR
* have etiologies of diffuse intrinsic pontine glioma, atypical teratoid rhabdoid tumor, or any tumor with cerebral or spinal metastases (these patients' clinical course and survival are highly unpredictable); OR
* are not expected to survive for 6 months; OR
* are unable or unwilling to participate in the study and with the neuropsychological exam; OR
* due to limitations of neuropsychological testing, blind and deaf children will be excluded. Children for whom English is not their primary language will be included if they have attended 1 or more years of English language based schooling.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric, school-aged patients presenting with a first time diagnosis of hydrocephalus.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Association between ventricle size and neuropsychological outcome | 6 months after initial surgical treatment for hydrocephalus
  Ventricle size, measured as fronto-occipital horn ratio (FOR), as well as neuropsychological outcomes at 6 months post-surgical intervention for initial treatment of hydrocephalus will be compared.

SECONDARY OUTCOMES:
Quality of life | 6 months after initial surgical treatment for hydrocephalus
  The Hydrocephalus Outcome Questionnaire (HOQ) will be administered at approximately 6 months. The HOQ is a validated measure of quality of life specific to the pediatric hydrocephalus population.
Academic Performance | 6 months after initial surgical treatment for hydrocephalus
  Parents will be asked to provide a picture of their child's current academic performance. If available, the child's most recent grade point average (GPA) will be obtained.
Presence of additional required hydrocephalus related surgeries | 6 months after initial surgical treatment for hydrocephalus
  Shunt and ETV revisions or infections will be examined for any correlations with cognitive neuropsychological testing at 6 months from the initial surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Riva-Cambrin, MD, MSc, Study Chair — Alberta Children's Hospital; Richard Holubkov, Ph.D., Principal Investigator — University of Utah
Locations (8):
- United States (7):
  - Children's Hospital of Alabama, University of Alabama, Birmingham, Alabama
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Sick Children's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hydrocephalus Clinical Research Network website — http://hcrn.org